CLINICAL TRIAL: NCT02673580
Title: Tele-patient-reported Outcomes (telePRO) in Clinical Practice - Effect of Patient-initiated Versus Fixed Interval telePRO Based Outpatient Follow-up
Brief Title: Tele-patient-reported Outcomes (telePRO) in Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TELEPRO
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2017-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

ARMS (2):
- Open Access telePRO (Other): Intervention: In open access, contact to the outpatient clinic is initiated by the patient by filling in a PRO questionnaire.
  Interventions: Other: Open Access telePRO
- Standard telePRO (Other): No intervention: In standard telePRO, outpatient follow-up activity is determined by a clinician and patients receive a questionnaire at fixed intervals.
  Interventions: Other: Standard telePRO

INTERVENTIONS:
Other: Open Access telePRO — In open access, contacts to the outpatient clinic are initiated solely by the patient. Contacts may be in the form of a PRO assessment like in standard telePRO, but at a time decided by the patient via the Danish National Health website "Sundhed.dk".
  Arms: Open Access telePRO
Other: Standard telePRO — Standard care: fixed interval telePRO follow-up. Patients receive a questionnaire with individually pre-specified intervals.
  Arms: Standard telePRO

SUMMARY:
The aim of this study is to compare quality of care and patient experiences in two outpatients follow-up activities: 1) Standard telePRO (fixed interval telePRO follow-up) and 2) Open Access telePRO (patient-initiated telePRO follow-up)

DETAILED DESCRIPTION:
The traditional system of routine outpatient follow-up of chronic disease in secondary care may involve a waste of resources if patients are well. The use of patient-reported outcomes (PRO) could support more flexible, cost-saving follow-up activities. AmbuFlex is a PRO system used in outpatient follow-up in the Central Denmark Region. PRO questionnaires are sent to patients at fixed intervals. The clinicians use the PRO data to decide whether a patient needs a visit or not (standard telePRO). PRO may make patients become more involved in their own care pathway, which may improve their self-management. Better self-management may also be achieved by letting patients initiate contact. The aim of this study is to obtain data on the effects of patient-initiated follow-up (open access telePRO) on resource utilisation, quality of care, and the patient perspective.

ELIGIBILITY:
Inclusion Criteria:

* Males and females from Age 15 years
* Diagnosis of epilepsy
* Referred to standard telePRO by a clinician
* Access to internet (web-responders in standard telePRO)
* Can speak and understand Danish

Exclusion Criteria:

* Paper responders
* Referred to telePRO proxy questionnaire

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of contacts | 18 months
  Number of contacts includes all contacts with the outpatient clinic in the study follow-up period

SECONDARY OUTCOMES:
General health will be assessed by items from the SF-36 questionnaire | 18 months
  General health will be measured at baseline and after 18 months.
Well-being wil be assessed by the WHO-5 Well-being Index | 18 months
  Well-being will be measured at baseline and after 18 months.
Mortality | 18 months
  Mortality will be measured after 18 months.
Number of seizures | 18 months
  Difference number of seizures (start - end) and will be measured at baseline and after 18 months.
Side effects | 18 months
  Side effects will be measured at baseline and after 18 months.
Health literacy will be assessed by The Health Literacy Questionnaire (sub scale 4, 6, and 9) | 18 months
  Health literacy will be measured at baseline and after 18 months.
Self-efficacy will be assessed by The General Self-Efficacy Scale | 18 months
  Self-efficacy will be measured at baseline and after 18 months.
Confidence will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 18 months
  Confidence will be measured at baseline and after 18 months.
Safety will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 18 months
  Safety will be measured at baseline and after 18 months.
Satisfaction will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 18 months
  Satisfaction will be measured at baseline and after 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henrik Hjollund, Professor, Study Director — Regional Hospital West Jutland
Locations (1):
- Regional Hospital West Jutland, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schougaard LMV, Mejdahl CT, Christensen J, Lomborg K, Maindal HT, de Thurah A, Hjollund NH. Patient-initiated versus fixed-interval patient-reported outcome-based follow-up in outpatients with epilepsy: a pragmatic randomized controlled trial. J Patient Rep Outcomes. 2019 Sep 13;3(1):61. doi: 10.1186/s41687-019-0151-0. PMID 31520247
- [Derived] Schougaard LM, Mejdahl CT, Petersen KH, Jessen A, de Thurah A, Sidenius P, Lomborg K, Hjollund NH. Effect of patient-initiated versus fixed-interval telePRO-based outpatient follow-up: study protocol for a pragmatic randomised controlled study. BMC Health Serv Res. 2017 Jan 26;17(1):83. doi: 10.1186/s12913-017-2015-8. PMID 28122609